CLINICAL TRIAL: NCT06734559
Title: Evaluation of the Effect of Acute Apical Periodontitis on Masseter Muscle With Elastography: A Case-control Study
Brief Title: Assessment of Masseter Muscle With Ultrasonography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Nezif Celik, assistant professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRÜ-DHF-END-NC-01
Record Dates: First submitted 2024-11-28; First posted 2024-12-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Acute Apical Periodontitis of Pulpal Origin
Keywords: pain; masseter; muscle; ultrasonography; teeth
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: two groups with control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound group (Active Comparator): Apical periodontitis' is a general term used to describe the periapical inflammatory process that occurs in response to the presence of micro-organisms and other irritants within the root canal system of a tooth. The length and mass of the masseter muscle will be measured on the first and 28th day of root canal treatment in patients with acute apical periodontitis..
  Interventions: Diagnostic Test: Patients who have not antibiotic treatment for acute apical periodontitis in the last month and have not taken any anti-inflammatory medication in the past 24 hours.
- sham group (Sham Comparator): Masseter muscle length and weight will be measured on the first and 28th day.
  Interventions: Other: patients who have not acute apical periodontitis

INTERVENTIONS:
Diagnostic Test: Patients who have not antibiotic treatment for acute apical periodontitis in the last month and have not taken any anti-inflammatory medication in the past 24 hours. — Patients with acute apical periodontitis will first have masseter muscle measurements in the relevant area and then the decayed tooth will be treated with calcium hydroxide for 14 days. Then the dressing will be applied with calcium hydroxide again. At the end of 28 days, the patient will be measured again by ultrasonography and the initial and final data will be compared.
  Arms: ultrasound group
Other: patients who have not acute apical periodontitis — Masseter measurements will be made from day 1 to day 28 in healthy subjects without acute apical periodontitis.
  Arms: sham group

SUMMARY:
In teeth that remain decayed for a long time, the muscles in that area atrophy because the patient cannot use the decayed area much. As a result, muscle length and mass decrease. To compare the amount of this reduction before and after treatment with ultrasound and to treat accordingly

DETAILED DESCRIPTION:
Material and method Clinical examination Apical periodontitis is inflammation of the periodontium at the entry portals of the root canal system. Typically, the lesion is found at the root apex, but it can occur at various levels along the root surface, and lesions can also develop in the lateral and furcal regions Acute apical periodontitis (AAP) is characterized by acute clinical symptoms (pain with the teeth in occlusion, tenderness to percussion or palpation in the periapical region, intrasulcular/intracanal pus drainage and swelling) but no evidence of periapical radiolucency except for mild widening of the periodontal ligament.

Patients will be selected from patients who apply to the Department of Endodontics, Faculty of Dentistry, Harran University, as a result of clinical and radiological examinations for acute apical periodontitis cases. After the patients are informed about the treatments to be performed, ultrasound measurements will be performed on the patients. Ultrasound(USG) imaging procedures will be performed by a single operator. Data will be recorded. Then, under local anesthesia and rubber dam isolation, the relevant tooth will be opened with round (Intensiv212) and Endo-Z (Dentsply-Maillefer) access cavities. Then, the canal length will be determined using 10-K (Dentsply-Maillefer) files and Propex Pixi (Dentsply Maillefer, Ballaigues, Switzerland). As expansion procedures, final shaping will be performed with F2 files using Protaper universal (Dentsply Maillefer, Ballaigues, Switzerland). The canals will be irrigated with 2 ml sodium hypochlorite at each file change. final irrigation will be done with 5ml 17% EDTA (Ethylenediaminetetraacetic acid), 2.5ml DW (distilled water) and 5.25% NaOCl (sodium hypochlorite). Then, after the canals are dried, they will be filled with calcium hydroxide and kept for 14 days with glass ionomer filling. At the end of this period, the patients will be called back, the necessary checks will be done, the canals will be washed again and kept for another 14 days with calcium hydroxide. At the end of the total of 28 days, the measurements will be repeated with a second ultrasound from the patients whose symptoms have completely disappeared and before and after comparisons will be made.

USG imaging In USG evaluation, LOGIQ P9 XDclear (GE HealthCare, USA) Masseter muscle thickness measurements will assume that the part with the highest repeatability is the middle part of the mediolateral line along the mandibular ramus. Therefore, when making measurements, the "L 3-12 RS (3-12 MHz)" linear probe will be placed approximately from the region corresponding to the middle of the mediolateral line along the mandibular ramus, perpendicular to the fibers of the masseter muscle, and parallel to the long axis of the corpus mandibula, in the middle between the zygomatic arch and the gonial angle, close to the occlusal plane, which is the thickest part of the masseter muscle.

Muscle thickness was defined as the maximum distance between the inner and outer fascia. Shear wave elastography (SWE) method will be used in ultrasonographic elastography examinations of muscles. In this study, the value recorded as Young's modulus will be defined as hardness and kPa units will be used.

Masseter Muscle SWE Examination For each participant, the stiffness values of the muscles at rest and at maximum contraction will be calculated for the right and left masseter muscles. The probe will be placed at the widest part in the middle of the muscle belly, perpendicular to the long axis of the masseter muscle. In the second method, the probe will be placed at the widest part in the middle of the muscle, parallel to the long axis of the masseter muscle.

In both methods, the middle part of the masseter muscle will be determined as the most prominent part when the participant bites in the B-Mode images. Then, the width of the region to be examined will be adjusted and the "Elasto" mode will be selected and the SWE system will be activated.

With the activation of the SWE system, the screen will be divided into right and left sections, where the routine grayscale image will be displayed on the left and the elastography image will be displayed on the right. Then, three consecutive elastography images will be obtained and a 10 cm2 circular region of interest (ROI) will be placed at the center of the examined muscle tissue in each image. After three measurements are taken in this way, the average of the measurements will be taken as the stiffness value of the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Having acute apical periodontitis
* Presence of at least four occlusal units in the posterior teeth (a pair of premolars in occlusion was counted as one unit, and a pair of molars in occlusion was counted as two units)
* over the age of 18
* Having no maxillofacial pathology or systemic disease
* Having no TMJ or masticatory muscle disorders
* People without complaints of dysphonia.
* Having no any muscle diseases

Exclusion Criteria:

* Having any systemic disease
* Using any type of drug
* Having less than 20 teeth
* Having prosthetic restoration (Single crowns, fixed dental prostheses, removable dental prostheses)
* Having implant restoration
* Have had periodontal treatment in the last one year
* Having a painful tooth (pulpitis)
* Pregnancy
* Smoking
* Unilateral edentulous patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
The thickness and length of the masseter muscle | first week
  Masseter muscle thickness measurements will made on the screen at the same time, with the help of the distance measurement feature of the USG device, over images of the muscles at rest and maximum contraction. masseter muscle thickness will be measured in millimeters (mm).
Masseter muscle stiffness | first week
  Masseter muscle stiffness will be measured in kilopascals (Kpa)

SECONDARY OUTCOMES:
The thickness and length of the masseter muscle | four weeks
  Masseter muscle thickness measurements will made on the screen at the same time, with the help of the distance measurement feature of the USG device, over images of the muscles at rest and maximum contraction. masseter muscle thickness will be measured in millimeters (mm).
Masseter muscle stiffness | four weeks
  Masseter muscle stiffness will be measured in kilopascals (Kpa)

CONTACTS AND LOCATIONS:
Overall Officials: nezif çelik, PhD, Study Director — HARRAN UNİVERSTY DENTİSTRY FACULTY; mehmet EMİN DOĞAN, PhD, Principal Investigator — HARRAN UNİVERSTY DENTİSTRY FACULTY
Locations (2):
- Turkey (Türkiye) (2):
  - Harran University, Sanliurfa, Haliliye
  - Nezif Çelik, Karaköprü, Şanlıurfa

IPD SHARING:
Plan to Share IPD: No